CLINICAL TRIAL: NCT03599999
Title: Study of Adverse Effects Occuring in Patients Receiving an Antibiotic Treatment With Temocillin
Acronym: Témocilline
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0003
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Bacterial Infection With One or More Extended Spectrum Betalactamases Remaining Susceptible to Temocillin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adverse events detection — type of adverse events detected during treatment with Temocillin and imputed to Temocillin

SUMMARY:
The Temocillin prescription frequency may be increased in order to reduce the use of carbapenems to reduce the progressive increase in carbapenem resistance observed in recent years. The investigators wish to study the responsibility of Temocillin in the occurrence of adverse effects in patients in the hospital of Amiens receiving a treatment containing this molecule.

DETAILED DESCRIPTION:
The study "Continuous versus intermittent infusion of temocillin, a directed spectrum penicillin for intensive care patients with nosocomial pneumoniae: stability, compatibility, population pharmacokinetic studies and breakpoint selection, R. De Jongh, et al, 2007 ", the author states that no adverse effects were found following injection of Temocillin. In the study "Temocillin use in England: clinical and microbiological efficacies in infections caused by extentedspectrum and / or derepressed AmpC β-lactamase-producing Enterobacteriaceae, I. Balakrishnan, et al, 2011, the author faced two cases of Clostridium difficile with a positive toxin test. The first patient received three doses of Amoxicillin / clavulanic acid followed by one week's treatment with Temocillin. This one has developed Clostridium difficile diarrhea on the last day of antibiotic treatment. The second patient did not not received Temocillin in the 6 weeks prior to diarrhea but received 8 days of Meropenem just before this diarrhea. In all cases, Temocillin can not be clearly attributed to this adverse effect and no patient developed pseudomembranous colitis.

ELIGIBILITY:
Inclusion Criteria:

* documented bacterial infection with one or more extended spectrum betalactamases remaining susceptible to Temocillin

Exclusion Criteria:

* History of hypersensitivity to betalactamines (rash,…)
* Patient participating in another biomedical research on a drug to avoid the risk of interactions drug
* Grafted patient
* Immunocompromised patient
* Dialysis patient (except hemodialysis patient and dialysis patient peritoneal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This concerns patients over the age of 18 years old with documented bacterial infection with one or more extended spectrum betalactamases remaining susceptible to Temocillin.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
number and type of adverse events detected during treatment with Temocillin and imputed to Temocillin | 7 days after the end of treatment
  Each reported case will be, first, analyzed by the principal investigator (an infectiologist), who will also be responsible for collecting information to fill out the data collection sheets and, secondarily, by the CRPV d'Amiens, which will bring its expertise in particular to define the imputability of Temocillin to the undesirable effect detected.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France